CLINICAL TRIAL: NCT00344539
Title: Phase I Study of the Safety and Immunogenicity of AMA1-C1/Alhydrogel® + CPG 7909, an Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria
Brief Title: AMA1-C1/Alhydrogel + CpG 7909 for Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-075
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-03

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: asexual blood stage vaccine, Plasmodium falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- B (Experimental): 80 mcg AMA1-C1/Alhydrogel® with 368 mcg Aluminum and 500 mg CPG 7909.
  Interventions: Biological: AMA1-C1/Alhydrogel®; Biological: CPG 7909 Oligodeoxynucleotide (VaxImmune®)
- C (Experimental): 80 mcg AMA1-C1/Alhydrogel® with 368 mcg Aluminum alone.
  Interventions: Biological: AMA1-C1/Alhydrogel®
- A (Experimental): 20 mcg AMA1-C1/Alhydrogel® with 377 mcg Aluminum and 500 mg CPG 7909.
  Interventions: Biological: AMA1-C1/Alhydrogel®; Biological: CPG 7909 Oligodeoxynucleotide (VaxImmune®)

INTERVENTIONS:
Biological: AMA1-C1/Alhydrogel® — AMA1-C1/Alhydrogel malaria vaccine, cloudy suspension, 0.5 mL dose containing up to equivalent of 377 mcg of aluminum as Alhydrogel® (800 mcg of aluminum hydroxide gel per dose) onto which 20 mcg or 80 mcg of recombinant AMA1-C1 is bound. Dosages: 20 mcg and 80 mcg administered via the deltoid muscle by IM injection
Biological: CPG 7909 Oligodeoxynucleotide (VaxImmune®) — CPG 7909 is an investigational agent and is supplied in sterile vials at 10mg/mL in phosphate buffered saline for intramuscular administration. Dosage 500 mcg.
  Arms: A; B

SUMMARY:
The purpose of this study is to test an experimental malaria vaccine in about 75 healthy adults, 18-45 years of age. The study will also test an experimental adjuvant which is a material added to a vaccine to help the body make more defense cells. The body's immune response (response to foreign substances) and the safety of the vaccine will be tested. All subjects will receive 3 doses of vaccine on days 0, 28, and 56 and doses may increase during the study. Participation in the study is expected to be up to 323 days and includes 16 visits. Study procedures include medical history, physical exams, urine and blood testing.

DETAILED DESCRIPTION:
This phase I, dose escalating study will evaluate the safety and immunogenicity of the experimental malaria vaccine AMA1-C1/Alhydrogel®, and the ability of the TLR-9 agonist CPG 7909 oligodeoxynucleotide (ODN) to augment antibody responses to the vaccine and alter the Th1/Th2 bias. The vaccine preparations to be studied contain an equal mixture of AMA1 from two different clones of Plasmodium falciparum (FVO and 3D7). Subjects will be randomly assigned to receive Alydrogel® formulated vaccine with or without CPG 7909 in a point of use formulation. The study will be conducted at the University of Rochester Vaccine and Treatment Evaluation Unit. Subjects for this study will be healthy adults between the ages of 18 and 45 years with no history of malaria or of recent travel to malaria-endemic areas. Subjects will be enrolled in three consecutive dose-escalation cohorts with review by a Safety Monitoring Committee between cohorts. Subjects will receive 3 vaccinations with the AMA1-C1/Alhydrogel® vaccine formulated in Alhydrogel® with or without CPG 7909 adjuvant over 2 months (0, 1, 2 months) by intramuscular (IM) injection. Subjects will have multiple blood samples obtained over the next 6 months. The primary objective of the study is to assess the safety, reactogenicity of the AMA1-C1/Alhydrogel® + CPG 7909 vaccine. The secondary objectives of the study include the following: to demonstrate that the addition of CPG 7909 improves the immune responses to AMA1-FVO and AMA1-3D7, as compared to AMA1-C1/Alhydrogel® at day 70 (14 days after 3rd vaccination; to determine the dose of AMA1-C1/Alhydrogel® + CPG 7909 that generates the highest serum antibody levels of AMA-FVO and AMA1-3D7 at day 70; to assess and compare the duration of antibody responses to AMA1-FVO and AMA1-3D7 proteins by enzyme-linked immunosorbent assay (ELISA) over an 8 month period (6 months after 3rd vaccination); and to perform exploratory studies of B and T cell populations both before and after vaccination. The safety trial endpoints include the frequency and severity of local and systemic adverse events after each dose reported on the subject diary card (solicited adverse events) or reported by subjects spontaneously (unsolicited adverse events) and the presence of abnormal clinical laboratory tests after immunization in each group. The immunogenicity endpoints include the frequency and titer of vaccine induced neutralizing and binding antibody, and the presence and quantity of antigen-specific B cells and CD4 and CD8 T cells producing specified cytokines following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years, inclusive.
* Good general health as a result of review of medical history and/or clinical tests.
* Available for the duration of the trial (34 weeks).
* Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

* Pregnancy as determined by a positive urine Beta-hCG (if female) at any point during the study.
* Participant unwilling to use highly effective contraception methods (such as: abstinence, birth control pills or birth control patches or vaginal ring, diaphragm with spermicide, IUD (intrauterine device), condom with spermicide, progestin implant or injection, surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation), or a partner who has had a vasectomy) for the duration of the trial (if female).
* Currently lactating and breast-feeding (if female).
* Evidence of clinically significant immunosuppressive, neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
* Laboratory evidence of liver disease (aspartate aminotransferase greater than 1.25 times the upper limit of normal of the testing laboratory).
* Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory).
* Laboratory evidence of hematologic disease (absolute neutrophil count <1,500/cubic mm; hemoglobin < 0.9 times the lower limit of normal of the testing laboratory, by sex; or platelet count <140,000/cubic mm).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* Serologic evidence of infection with HIV-1, HBV, or HCV.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or while the study is ongoing.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of surgical splenectomy.
* Receipt of blood products within the past 6 months.
* Previous receipt of an investigational malaria vaccine.
* Receipt of antimalarial prophylaxis during the past 12 months.
* Prior malaria infection.
* Travel to a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* History of a known allergy to nickel.
* Pre-existing autoimmune or antibody mediated diseases including but not limited to: systemic lupus erythematosis, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia; or laboratory evidence of possible autoimmune disease determined by a positive anti-dsDNA titer, positive rheumatoid factor, proteinuria and/or a positive ANA.
* Chloroquine and related compounds within 12 weeks of study entry.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cellular immune response to vaccination. | Anti-AMA1 antibody will be measured by ELISA on Days 0, 14, 28, 42, 56, 70, 84, 140, and 236.
Serum antibody response to vaccination. | Day 70.
Safety: frequency of vaccine-associated adverse events, as classified by severity through active and passive surveillance. | Duration of study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Result] Mullen GE, Ellis RD, Miura K, Malkin E, Nolan C, Hay M, Fay MP, Saul A, Zhu D, Rausch K, Moretz S, Zhou H, Long CA, Miller LH, Treanor J. Phase 1 trial of AMA1-C1/Alhydrogel plus CPG 7909: an asexual blood-stage vaccine for Plasmodium falciparum malaria. PLoS One. 2008 Aug 13;3(8):e2940. doi: 10.1371/journal.pone.0002940. PMID 18698359